CLINICAL TRIAL: NCT03341910
Title: A Randomized, Double-Blind, Active-Controlled Study to Assess the Safety and Local Tolerability of DFD-03 (Tazarotene) Lotion, 0.1% Compared to Tazorac® (Tazarotene) Cream, 0.1% in the Topical Treatment of Acne Vulgaris for 12 Weeks
Brief Title: A Study to Assess the Safety and Local Tolerability of DFD-03 (Tazarotene) Lotion, 0.1% Compared to Tazorac® Cream, 0.1% in the Topical Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFD-03-CD-008
Record Dates: First submitted 2017-10-13; First posted 2017-11-14 (Actual); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DFD-03 Lotion, 0.1% (Experimental): DFD-03 Lotion, 0.1% to be applied twice daily approximately 12 hours apart, for 1 minute and rinsed off
  Interventions: Drug: DFD-03 Lotion, 0.1%
- Tazorac Cream, 0.1% (Active Comparator): Tazorac Cream, 0.1% to be applied once in the evening and left overnight for approximately 12 hours
  Interventions: Drug: Tazorac Cream, 0.1%
- Vehicle Lotion (Placebo Comparator): Vehicle Lotion to be applied twice daily for 1 minute and rinsed off
  Interventions: Drug: DFD-03 Vehicle Lotion 0%
- Vehicle Cream (Placebo Comparator): Vehicle Cream to be applied once in the evening and left overnight for approximately 12 hours
  Interventions: Drug: Tazorac Vehicle Cream 0%

INTERVENTIONS:
Drug: DFD-03 Lotion, 0.1% — DFD-03 Lotion will be applied to the face (avoiding areas around the eyes and mouth) twice daily, approximately 12 hours apart, and washed off after 1 minute.
  Other Names: Tazarotene Lotion, 0.1%
  Arms: DFD-03 Lotion, 0.1%
Drug: Tazorac Cream, 0.1% — Tazorac Cream will be applied to the face (avoiding areas around the eyes and mouth) once daily in the evening and left on overnight.
  Other Names: Tazarotene Cream, 0.1%
  Arms: Tazorac Cream, 0.1%
Drug: DFD-03 Vehicle Lotion 0% — Vehicle Lotion will be applied to the face (avoiding areas around the eyes and mouth) twice daily, approximately 12 hours apart, and washed off after 1 minute.
  Other Names: Vehicle Lotion 0%
  Arms: Vehicle Lotion
Drug: Tazorac Vehicle Cream 0% — Vehicle Cream will be applied to the face (avoiding areas around the eyes and mouth) once daily in the evening and left on overnight.
  Other Names: Vehicle Cream 0%
  Arms: Vehicle Cream

SUMMARY:
A study for Subjects with mild to moderate facial acne vulgaris. During the 12-week treatment period subjects randomized to DFD-03 Lotion or Vehicle Lotion will use the study drug twice daily. Subjects randomized to Tazorac Cream or Vehicle Cream will use the study drug once daily in the evening. Safety assessments will include the investigator's assessment of local cutaneous tolerance/application site reactions on the face, vital signs and adverse events.

DETAILED DESCRIPTION:
A study for Subjects with mild to moderate facial acne vulgaris. Subjects will be randomized to treatment with either DFD-03 (tazarotene) Lotion 0.1%, Tazorac (tazarotene) Cream, 0.1%, Vehicle Lotion or Vehicle Cream. During the 12-week treatment period subjects randomized to DFD-03 Lotion or Vehicle Lotion will use the study drug twice daily. Subjects randomized to Tazorac Cream or Vehicle Cream will use the study drug once daily in the evening. Subjects will be instructed to treat the entire face.

Safety assessments will include the investigator's assessment of local cutaneous tolerance/application site reactions on the face, vital signs and adverse events. Urine pregnancy tests will be performed for all female subjects. A physical examination will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 12 years of age. At selected site(s), a total of approximately eight subjects 9-11 years of age will be enrolled into the 2 arms of DFD-03 lotion group (active and vehicle).
2. A clinical diagnosis of facial acne vulgaris with a facial Investigator's Global Assessment (IGA) score of 2 (mild) to 3 (moderate) at Baseline. At selected site(s), up to twelve subjects with acne lesions on the chest and/or back (including shoulders) in addition to those on the face will treat their chest and/or back (including shoulders) in addition to their face.
3. Inflammatory lesion count (papules and pustules) of at least 20, non-inflammatory lesion count (closed and open comedones) of at least 25 on the face including the nose, and no more than 2 nodulocystic lesions. This criteria is not applicable to the 9-11 years age group as long as subjects have an IGA score of 2 (mild) to 3 (moderate) at Baseline.
4. Females, regardless of childbearing potential: Must have a negative urine pregnancy test and if sexually active, must be on or use an acceptable method of birth control.
5. Subjects agree not to use any product on the face during the entire course of study except for non-medicated, investigator-approved cleanser, sunscreen, face wash, and make-up as instructed by the investigator.
6. Subjects must be willing to comply with sun avoidance measures for the face, including use of investigator-approved sunscreen and/or hats, have limited sun exposure time, and have no tanning bed use.
7. Subject must be in good general health as determined by the investigator and supported by the medical history, physical examination and vital signs.

Exclusion Criteria:

1. Females who are pregnant or lactating or planning to become pregnant during the study period.
2. Treatment with the following products:

   Topical acne treatments or other topical facial medication in the 14 days prior to Baseline Systemic corticosteroids and systemic acne treatments in the 30 days prior to Baseline Systemic retinoid use in the 180 days prior to Baseline Undertaken certain facial procedures such as chemical peel, laser treatment, photodynamic therapy, acne surgery, cryodestruction or chemodestruction, x-ray therapy, intralesional steroids, dermabrasion, or depilation (except eyebrow shaping) in 30 days prior to Baseline.

   Treatment with a medication or procedure that, in the opinion of the investigator, would put the subject at unacceptable risk for participation in the study or may interfere with evaluations in the study.

   Treatment with an investigational product or device in 30 days prior to Baseline.
3. Known allergic reaction to retinoids or tazarotene or any of the product ingredients.
4. Presence of any facial skin disease or condition that would interfere with the study or place the subject at unacceptable risk including sunburn, rosacea, seborrheic dermatitis, perioral dermatitis, lupus, dermatomyositis, psoriasis, eczema, squamous cell carcinoma, acneiform eruptions caused by medications, steroid acne, steroid folliculitis, bacterial folliculitis or any other facial disease or condition.
5. Subjects with a serious and or chronic medical condition such as chronic or active liver disease, renal impairment, heart disease, severe respiratory disease, rheumatoid arthritis, current malignancies, immunocompromised conditions, or any other disease that, in the opinion of the investigator, would interfere with the study or place the subject at unacceptable risk.
6. Subjects who have been treated for alcohol dependence or alcohol or drug abuse in the year.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas R. Sidgiddi, M.D., Study Director — Dr. Reddy's Laboratories Inc.
Locations (1):
- International Dermatology Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DFD-03 Vehicle Lotion: Vehicle Lotion to be applied twice daily for 1 minute and rinsed off
  DFD-03 Vehicle Lotion 0%: Vehicle Lotion will be applied to the face (avoiding areas around the eyes and mouth) twice daily, approximately 12 hours apart, and washed off after 1 minute.
- Tazorac Vehicle Cream: Vehicle Cream to be applied once in the evening and left overnight for approximately 12 hours
  Tazorac Vehicle Cream 0%: Vehicle Cream will be applied to the face (avoiding areas around the eyes and mouth) once daily in the evening and left on overnight.
Period: Overall Study
Arm/Group | DFD-03 Lotion, 0.1% | Tazorac Cream, 0.1% | DFD-03 Vehicle Lotion | Tazorac Vehicle Cream
Started | 54 | 49 | 26 | 26
Completed | 54 | 49 | 26 | 26
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population - All subjects who received study product and provided any post-baseline safety information.
Groups:
- Total: Total of all reporting groups
Arm/Group | DFD-03 Lotion, 0.1% | Tazorac Cream, 0.1% | DFD-03 Vehicle Lotion | Tazorac Vehicle Cream | Total
Number analyzed (Participants) | 54 | 49 | 26 | 26 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 13 | 10 | 9 | 52
  Between 18 and 65 years | 34 | 36 | 16 | 17 | 103
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (9.5) | 23.1 (8.9) | 22.0 (9.7) | 25.0 (10.5) | 22.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 12 | 12 | 76
  Male | 29 | 22 | 14 | 14 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 2 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 4 | 5 | 3 | 6 | 18
  White | 46 | 44 | 20 | 18 | 128
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 54 | 49 | 26 | 26 | 155

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event Occurences in DFD-03 Lotion Versus Tazorac Cream Groups
Description: Frequency count of treatment emergent adverse events will be compared between DFD-03 Lotion and Tazorac Cream groups.
Time Frame: Baseline to Week 12
Population: Safety Population - All subjects who received study product and provided any post baseline safety information.
Measure: Number; unit: Adverse Events
Arm/Group | DFD-03 Lotion, 0.1% | Tazorac Cream, 0.1% | DFD-03 Vehicle Lotion | Tazorac Vehicle Cream
Number analyzed (Participants) | 54 | 49 | 26 | 26
Adverse Events | 73 | 81 | 14 | 15

ADVERSE EVENTS:
Time Frame: Adverse events were collected from treatment initiation until study product treatment discontinuation (approximately 12 weeks).
Description: Adverse events were collected from treatment initiation until study product treatment discontinuation (approximately 12 weeks). Spontaneously reported SAEs, which were reported up to 30 days after discontinuing study product use (approximately 4 months).
Groups:
- DFD-03 Lotion, 0.1%: DFD-03 Lotion, 0.1% was applied twice daily approximately 12 hours apart, for 1 minute and rinsed off
  DFD-03 Lotion, 0.1%: DFD-03 Lotion was applied to the face (avoiding areas around the eyes and mouth) twice daily, approximately 12 hours apart, and washed off after 1 minute.
- Tazorac Cream, 0.1%: Tazorac Cream, 0.1% was applied once in the evening and left overnight for approximately 12 hours
  Tazorac Cream, 0.1%: Tazorac Cream was applied to the face (avoiding areas around the eyes and mouth) once daily in the evening and left on overnight.
- Vehicle Lotion: Vehicle Lotion was applied twice daily for 1 minute and rinsed off
  DFD-03 Vehicle Lotion 0%: Vehicle Lotion was applied to the face (avoiding areas around the eyes and mouth) twice daily, approximately 12 hours apart, and washed off after 1 minute.
- Vehicle Cream: Vehicle Cream was applied once in the evening and left overnight for approximately 12 hours
  Tazorac Vehicle Cream 0%: Vehicle Cream was applied to the face (avoiding areas around the eyes and mouth) once daily in the evening and left on overnight.
Arm/Group | DFD-03 Lotion, 0.1% | Tazorac Cream, 0.1% | Vehicle Lotion | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/49 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/49 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 22/54 | 26/49 | 9/26 | 11/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD-03 Lotion, 0.1% (N=54) | Tazorac Cream, 0.1% (N=49) | Vehicle Lotion (N=26) | Vehicle Cream (N=26)
Application site dryness (General disorders) | 18 (18) | 17 (17) | 2 (2) | 3 (3)
Application site exfoliation (General disorders) | 14 (14) | 12 (12) | 2 (2) | 3 (3)
Application Site Pain (General disorders) | 14 (14) | 13 (13) | 1 (1) | 1 (1)
Application Site Erythema (General disorders) | 8 (8) | 9 (9) | 1 (1) | 3 (3)
Application Site Pruritus (General disorders) | 6 (6) | 3 (3) | 2 (2) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (5) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT03341910/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT03341910/SAP_001.pdf